CLINICAL TRIAL: NCT04893226
Title: Time-Restricted Feeding Intervention in Metabolically-Unhealthy Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Pendergast (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Julie Pendergast, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIO-21-TRF; 1R01DK124774-01A1 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Syndrome; Postmenopausal Symptoms
Keywords: postmenopause; weight; metabolic risk; glucose; body composition; lipid; sleep; prediabetes; fasting; circadian; inflammation
MeSH Terms: conditions — Metabolic Syndrome; Body Weight; Prediabetic State; Fasting; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in this group will have baseline and post-study data collected, including food timing, activity/sleep data, and metabolic parameters (OGTT, body composition, anthropometric measurements, lipid panel, inflammatory markers). There will be no intervention.
- Time-Restricted Feeding (TRF) Group (Experimental): Participants in this group will have baseline and post-study data collected, including food timing, activity/sleep data, and metabolic parameters (OGTT, body composition, anthropometric measurements, lipid panel, inflammatory markers). Subjects in this group will be educated about the health benefits of time-restricted feeding (TRF). Then each subject in the TRF group will self-select a 10-h window during which she will consume all daily calories for 16 weeks.
  Interventions: Behavioral: Time-Restricted Feeding (TRF)

INTERVENTIONS:
Behavioral: Time-Restricted Feeding (TRF) — Subjects will be educated about the health benefits of time-restricted feeding (TRF). Each subject in the TRF group will self-select a 10 hour (10h +/- 1hr) window aligned with their active phase during which they will consume all daily calories. Subjects will text the time of their first and last daily meals for the duration of the study.
  Arms: Time-Restricted Feeding (TRF) Group

SUMMARY:
This is a randomized, parallel two-arm clinical trial design to study the efficacy of time-restricted feeding on metabolic risk in postmenopausal women, who may be particularly vulnerable to disruption of circadian eating rhythms and the associated metabolic dysfunction. It is hypothesized that time-restricted feeding will improve insulin sensitivity, glucose tolerance, body weight, and other metabolic parameters in metabolically-unhealthy postmenopausal women.

DETAILED DESCRIPTION:
This is a randomized, parallel two-arm clinical trial design to study the efficacy of time-restricted feeding (TRF) on metabolic risk in postmenopausal women. Data will be collected for 18 weeks. Baseline food timing, activity/sleep, and metabolic parameter (OGTT, body composition, anthropometric measurements, lipid panel, inflammatory markers) data will be collected in the first two weeks (baseline). Subjects will then be randomized to the TRF intervention or no TRF for 16 weeks. Subjects in the TRF group will be educated about the health benefits of TRF. Then each subject in the TRF group will self-select a 10-h window and consume all daily calories during this time frame. Subjects in both the TRF and no TRF groups will text the time of their first and last daily meals for the duration of the study. At the end of the 16-week TRF intervention or no TRF, metabolic and anthropometric measurements will be collected.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* age 45-65 years
* prediabetic or have at least 2 features of metabolic syndrome

Exclusion Criteria:

* on hormone therapy
* diabetes
* heart disease
* alcohol consumption of >2 drinks per day
* significant circadian disruption
* having care-taking responsibilities that significantly affect sleep
* shift work or irregular lifestyle
* uncontrolled sleep apnea or other uncontrolled sleep disorder
* extreme early or late chronotypes
* significant psychiatric disorders
* taking ADHD medications
* diagnosed dysregulated eating behaviors
* smoking >5 cigarettes/day or 30 pack-year history
* participating in formal weight loss program
* not weight stable

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity | 18 weeks (baseline and post-intervention)
  Matsuda index will be assessed by the oral glucose tolerance test (OGTT).
Change in Body Mass Index | 18 weeks (baseline and post-intervention)
  Body mass index will be calculated from height and weight.
Change in Triglycerides | 18 weeks (baseline and post-intervention)
  Triglycerides will be measured from fasting blood

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | 18 weeks (baseline and post-intervention)
  HbA1c is a measure of the proportion of glycated hemoglobin in blood.
Change in C-Reactive Protein | 18 weeks (baseline and post-intervention)
  CRP will be measured from blood samples.
Change in Mid-sleep | 18 weeks (baseline and post-intervention)
  Mid-sleep is a single outcome calculated using both actigraphy and sleep log information.
Change in Sleep Fragmentation Index | 18 weeks (baseline and post-intervention)
  Sleep fragmentation index, a measure of sleep quality, will be assessed from actigraphy data.

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Pendergast, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No